CLINICAL TRIAL: NCT00124657
Title: A Phase I/II Trial of a New Tyrosine Kinase Inhibitor (Tarceva; Erlotinib Hydrochloride; OSI-774) During and After Radiotherapy in the Treatment of Patients With Newly Diagnosed High Grade Glioma and Unfavorable Low-Grade Glioma
Brief Title: Erlotinib and Radiation Therapy in Treating Young Patients With Newly Diagnosed Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Rady Children's Hospital, San Diego (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJHG04
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; adult mixed glioma; childhood mixed glioma; untreated childhood cerebellar astrocytoma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebral astrocytoma; childhood oligodendroglioma; childhood spinal cord neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Spinal Cord Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with High-Grade/Low-Grade Glioma (Experimental): Patients with newly diagnosed high-grade glioma (excluding those originating in the brain stem) and unfavorable low-grade glioma who are ≥ 3 years and <26 years of age. Patients receiving enzyme-inducing anticonvulsants (EIACs) are not eligible for this study. Patients with spinal cord tumors will be eligible for the Phase I and Phase II component of this study, but they will not be taken into consideration to estimate PFS in the Phase II component of this trial because of their notoriously worse prognosis. Patients receive erlotinib hydrochloride.
  Interventions: Drug: Erlotinib hydrochloride

INTERVENTIONS:
Drug: Erlotinib hydrochloride — This study has 2 components: a Phase I component which estimated the MTD and DLT(s) of erlotinib given once a day during and after conventionally fractionated RT for a period of 8 weeks (DLT-evaluation period), followed by continuous administration of this medication for up to 3 years; and a Phase II component where erlotinib will be given at the MTD during and after RT for 2 years. The recommended dose of erlotinib for the Phase II component of the current study is 120mg/m2 per day (maximum dose of 200mg per day).
  Other Names: Tarceva; OSI-774; NSC#718781

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It may also make tumor cells more sensitive to radiation therapy. Giving radiation therapy together with erlotinib may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of erlotinib when given together with radiation therapy and to see how well they work in treating young patients with newly diagnosed glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicity of erlotinib when administered during and after radiotherapy in young patients with newly diagnosed high-grade glioma and unfavorable low-grade glioma.
* Determine the 1- and 2-year progression-free survival of patients treated with this regimen.

Secondary

* Determine the toxic effects of this regimen in these patients.
* Correlate genetic abnormalities in epidermal growth factor receptor (EGFR) and components of downstream pathways with treatment response in patients treated with this regimen.
* Determine the ability of erlotinib to inhibit EGFR signaling in patients with high-grade glioma who require second surgery.
* Determine the pharmacokinetics of erlotinib and its metabolites in these patients.
* Correlate plasma and cerebrospinal fluid levels of vascular endothelial growth factor and basic fibroblast growth factor with tumor response in patients treated with this regimen.
* Correlate irradiation dosimetry with patterns of failure, standard and investigational imaging, and toxicity in patients treated with this regimen.

OUTLINE: This is a phase I dose-escalation study of erlotinib followed by a phase II study.

* Phase I: Patients undergo radiotherapy once daily, 5 days week, for approximately 6½ weeks. Beginning on the first day of radiotherapy, patients receive oral erlotinib once daily for up to 2 years.

Cohorts of patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined.

* Phase II: Patients will receive erlotinib as in phase I at the MTD and undergo radiotherapy as in phase I.

PROJECTED ACCRUAL: A total of 75-80 patients (15-20 for the phase I portion and 60 for the phase II portion) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of high-grade glioma of 1 of the following types:

  * Unfavorable low-grade glioma

    * Gliomatosis cerebri or bithalamic involvement
  * Histologically confirmed high-grade glioma (WHO grade III or IV) of 1 of the following subtypes:

    * Anaplastic astrocytoma
    * Anaplastic oligodendroglioma
    * Anaplastic oligoastrocytoma
    * Anaplastic ganglioglioma
    * Pleomorphic xanthoastrocytoma with anaplastic features
    * Malignant glioneuronal tumor
    * Glioblastoma multiforme
    * Gliosarcoma
* Newly diagnosed disease
* Intracranial or spinal cord tumors allowed

PATIENT CHARACTERISTICS:

Age

* 3 to 21

Performance status

* Karnofsky 40-100% (age 17 to 21 years) OR
* Lansky 40-100% (age 3 to 16 years)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 8 g/dL (transfusion allowed)

Hepatic

* Bilirubin < 1.5 times upper limit of normal (ULN)
* SGPT < 5 times ULN
* Albumin ≥ 2 g/dL

Renal

* Creatinine < 2 times normal OR
* Glomerular filtration rate > 70 mL/min

Cardiovascular

* No significant cardiovascular problem

Pulmonary

* No significant pulmonary problem

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No uncontrolled infection
* No significant medical illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior or concurrent biologic agents

Chemotherapy

* No prior or concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* No more than 42 days since prior surgery

Other

* No other prior or concurrent anticancer or experimental treatment

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2005-03; Primary Completion 2012-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Broniscer, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - University of California San Diego, San Diego, California
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall accrual included 62 unique subjects. Five subjects participated in both Phase I and Phase II. Phase I enrolled 23 (03/2005-06/2007). Phase II enrolled an additional 39 participants (08/2007-11/2010) plus 5 carried over from Phase I for a total of 44. One of the 39 accrued to Phase II was enrolled at Rady Children's Hospital.
Pre-assignment Details: Participants had newly diagnosed high-grade glioma (except those originating in the brain stem) and unfavorable low-grade glioma and were ≥ 3 and ≤21 years of age. Participants receiving enzyme-inducing anticonvulsants (EIACs) were not eligible for this study. Patients with spinal cord tumors were eligible for the Phase II component of this study.
Groups:
- Phase I Only: 18 participants were enrolled on the Phase I portion of the trial only.
- Phase I and Phase II: 5 patients participated in both the Phase I portion and the Phase II portion of the study.
- Phase II Only: 39 participants were enrolled on the Phase II portion of the trial only.
Period: Overall Study
Arm/Group | Phase I Only | Phase I and Phase II | Phase II Only
Started | 18 | 5 | 39
Completed | 2 | 0 | 7
Not Completed | 16 | 5 | 32
Not completed — Toxicity | 0 | 0 | 1
Not completed — Non-compliance | 1 | 0 | 4
Not completed — Progressive disease | 14 | 5 | 27
Not completed — Intercurrent illness | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Only | Phase I and Phase II | Phase II Only | Total
Number analyzed (Participants) | 18 | 5 | 39 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.49 (4.31) | 11.47 (6.05) | 10.55 (4.85) | 11.12 (4.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 23 | 33
  Male | 10 | 3 | 16 | 29
Diagnosis [Number; unit: participants]
  Anaplastic astrocytoma (AA) | 7 | 1 | 19 | 27
  Glioblastoma multiforme (GBM) | 8 | 4 | 17 | 29
  Anaplastic oligoastrocytoma | 2 | 0 | 1 | 3
  Anaplastic ganglioglioma | 1 | 0 | 0 | 1
  Unfavorable fibrillary astrocytoma | 0 | 0 | 1 | 1
  Spinal GBM | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT)
Description: DLT was defined as any of the following toxicities attributable to erlotinib therapy: thrombocytopenia grade 3 and 4; neutropenia grade 4; or any grade 3 and 4 non-hematologic toxicity except for grade 3 diarrhea and grade 3 nausea and vomiting lasting ≤48 hours in participants not receiving optimal supportive therapy, grade 3 skin rash, which did not affect normal daily activities, grade 3 fever or nonneutropenic infection, grade 3 seizures, grade 3 weight gain or loss, and grade 3 transaminase elevation that returned to grade 1 or baseline within 7 days. After enrollment of the first 4 participants, grade 3 and 4 electrolyte abnormalities that resolved to ≤grade 2 within 7 days were excluded as DLT. Toxicities were graded according to the Common Terminology Criteria for Adverse Events version 3.0.
Time Frame: During the first 8 weeks of therapy
Population: 23 participants were enrolled on Phase I component; 22 were analyzed for DLT over 4 dose levels. 1 treated at dose level 120mg/m^2 was not assessable for DLT due to early tumor progression. 4 were treated before and 19 after the study was amended to exclude grade 3 and 4 electrolyte abnormalities that resolved to ≤ grade 2 within 7 days.
Measure: Number; unit: participants
Groups:
- 70 mg/m^2: Dose level 1 was 70 mg/m^2, range of actual dosage was 68-83 mg/m^2.
- 90 mg/m^2: Dose level 2 was 90 mg/m^2, range of actual dosage was 85-87.5 mg/m^2.
- 120 mg/m^2: Dose level 3 was 120 mg/m^2, range of actual dosage was 107-128 mg/m^2.
- 160 mg/m^2: Dose level 4 was 160 mg/m^2, range of actual dosage was 151.5-167 mg/m^2.
Arm/Group | 70 mg/m^2 | 90 mg/m^2 | 120 mg/m^2 | 160 mg/m^2
Number analyzed (Participants) | 7 | 3 | 6 | 6
participants | 0 | 0 | 1 | 2

2. Secondary Outcome: Cmax of Erlotinib and Its Metabolite OSI-420
Description: Although the calculated dose of erlotinib was rounded to the nearest 25 mg, the actual dosage administered to patients was within 12% of the prescribed dosage in all but 1 patient. The latter patient received erlotinib at the lowest dosage level and the actual dosage was 19% higher than the calculated dose.
Time Frame: After first dose of therapy, and Day 8 of therapy
Population: Pharmacokinetic variables were obtained in 17 patients enrolled on the Phase I portion of the study.
Measure: Median (Full Range); unit: mg/mL
Arm/Group | 70 mg/m^2 | 90 mg/m^2 | 120 mg/m^2 | 160 mg/m^2
Number analyzed (Participants) | 7 | 2 | 5 | 3
mg/mL
  Erlotinib, after first dose of therapy | 1.3 [0.94 to 2.2] | 1.6 [1.3 to 1.8] | 1.2 [0.5 to 2] | 1.8 [1.3 to 3]
  Erlotinib, Day 8 of therapy | 1.8 [1.7 to 2.8] | 1.3 [1.3 to 1.3] | 1.4 [1 to 3] | 2 [1.3 to 2.4]
  OSI-420, after first dose of therapy | 0.13 [0.05 to 0.2] | 0.16 [0.12 to 0.2] | 0.14 [0.1 to 0.3] | 0.32 [0.26 to 0.33]
  OSI-420, Day 8 of therapy | 0.25 [0.2 to 0.6] | 0.17 [0.17 to 0.17] | 0.3 [0.1 to 0.5] | 0.3 [0.3 to 0.3]

3. Secondary Outcome: Erlotinib Tmax
Description: as for outcome 2
Time Frame: After first dose of therapy
Population: Pharmacokinetic variables were obtained in 17 patients enrolled on the Phase I portion of the study.
Measure: Median (Full Range); unit: hours
Arm/Group | 70 mg/m^2 | 90 mg/m^2 | 120 mg/m^2 | 160 mg/m^2
Number analyzed (Participants) | 7 | 2 | 5 | 3
hours
  Erlotinib, after first dose of therapy | 4 [2.1 to 8.2] | 3.1 [2 to 4.1] | 2.2 [1 to 4] | 2.2 [2 to 2.5]
  Erlotinib, Day 8 of therapy | 2.1 [1 to 4.1] | 2.6 [1.2 to 4] | 1.75 [1.3 to 4] | 2.2 [1 to 4]

4. Secondary Outcome: AUC Time 0-infinite (AUCinf) of Erlotinib and Its Metabolite OSI-420
Description: as for outcome 2
Time Frame: After first dose of therapy, and Day 8 of therapy
Population: Pharmacokinetic variables were obtained in 17 patients enrolled on the Phase I portion of the study.
Measure: Median (Full Range); unit: mg*h/mL
Arm/Group | 70 mg/m^2 | 90 mg/m^2 | 120 mg/m^2 | 160 mg/m^2
Number analyzed (Participants) | 7 | 2 | 5 | 3
mg*h/mL
  Erlotinib, after first dose of therapy | 34.9 [23.1 to 52.6] | 23.9 [14.4 to 33.3] | 27.8 [18.9 to 28.8] | 37.1 [33.1 to 50.6]
  Erlotinib, Day 8 of therapy | 28.8 [21.8 to 30.9] | 21.2 [18.1 to 24.2] | 23.1 [11.8 to 51.2] | 35.5 [23.7 to 51]
  OSI-420, after first dose of therapy | 2.1 [1.2 to 3.3] | 1.9 [1.4 to 2.3] | 2.5 [1.7 to 2.7] | 4.2 [4.1 to 5.2]
  OSI-420, Day 8 of therapy | 3.3 [2 to 6.9] | 2.1 [1.7 to 2.4] | 2.8 [1.9 to 5.9] | 4.3 [3.8 to 6.1]

5. Secondary Outcome: Number of Positive Mutations of EGFR and Downstream Pathways
Description: Statistical analyses of genomic changes, expression profiles and validation studies should be considered in an exploratory and hypothesis-generating context.
  Fresh frozen tumor tissue was obtained at the time of tumor resection and diagnosis. DNA was extracted from formalin-fixed, paraffin-embedded tissue. The entire PTEN coding sequence (exons 1-9), exons 1, 9 and 20 of PIK3CA, and exons 17-24 of EGFR were evaluated using exon-specific PCR amplification, and immunohistochemistry was done. Tumor lesions were considered positive if >25% cells were immunoreactive.
Time Frame: Once at tumor resection and diagnosis
Population: Unstained slides were available for immunohistochemistry analysis in 21 of the 23 Phase I participants.
Measure: Number; unit: participants
Groups:
- Phase I: Phase I participants
Arm/Group | Phase I
Number analyzed (Participants) | 21
participants
  Positive for PTEN (R130*) | 1
  Positive PIK3CA (H1047R) | 1
  Positive EGFR kinase domain | 0

6. Primary Outcome: Maximum Tolerated Dose (MTD) of Erlotinib
Description: MTD was defined as the highest dosage level in which no more than one of six assessable participants experienced dose-limiting toxicities (DLT). The dosage of erlotinib was increased by approximately 30% in each dosage level starting at 80% of the MTD in adults with solid tumors. A traditional 3+3 dose escalation scheme was used to estimate the MTD.
Time Frame: During the first 8 weeks of therapy.
Population: 22 participants were analyzed for MTD over 4 dose levels. One of 23 enrolled participants was not evaluable due to early disease progression.
Measure: Number; unit: mg/m^2
Groups:
- Phase I: 22 participants were analyzed for MLT over 4 dose levels.
Arm/Group | Phase I
Number analyzed (Participants) | 22
mg/m^2 | 120

7. Primary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) distributions for the Phase II participants with anaplastic astrocytoma (AA) and glioblastoma multiforme (GBM) were calculated using Kaplan-Meier estimates (n=41). PFS was defined as the interval between treatment start and initial failure, including clinical or radiologic progression or death from any cause.
  PFS was not calculated for the other disease types.
Time Frame: 1 and 2 years after end of therapy
Population: Per protocol, 41 participants with either anaplastic astrocytoma or glioblastoma multiforme were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: years
Groups:
- Phase I AA: All participants with a diagnosis of anaplastic astrocytoma (AA) and treated on Phase I.
- Phase I GBM: All participants with a diagnosis of glioblastoma multiforme (GBM) and treated on Phase I.
- Phase II AA: Participants with a diagnosis of intracranial anaplastic astrocytoma (AA) treated with a combination of maximum safe surgical resection, local RT, and erlotinib.
- Phase II GBM: Participants with a diagnosis of intracranial glioblastoma multiforme (GBM) treated with a combination of maximum safe surgical resection, local RT, and erlotinib.
Arm/Group | Phase I AA | Phase I GBM | Phase II AA | Phase II GBM
Number analyzed (Participants) | 8 | 12 | 20 | 21
years
  1-year PFS | 0.75 (0.14) | 0.33 (0.12) | 0.45 (0.106) | 0.19 (0.077)
  2-year PFS | NA (NA) — 2-year PFS was not done by diagnosis group for Phase I participants. | NA (NA) — 2-year PFS was not done by diagnosis group for Phase I participants. | 0.15 (0.069) | 0.19 (0.077)
Statistical Analysis 1: Comparison: Phase I AA; 1-year progression-free survival (n=8); Test type: Superiority or Other; Kaplan-Meier = 0.75, 95% CI 2-sided [0.48 to 1.00], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Phase I GBM; 1-year progression-free survival (n=12); Test type: Superiority or Other; Kaplan-Meier = 0.33, 95% CI 2-sided [0.09 to 0.57], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Phase II AA; 1-year progression free survival (n=20); Test type: Superiority or Other; Kaplan-Meier = 0.45, 95% CI 2-sided [0.198 to 0.602], Standard Deviation 0.106
Statistical Analysis 4: Comparison: Phase II AA; 2-year progression free survival (n=20); Test type: Superiority or Other; Kaplan-Meier = 0.150, 95% CI 2-sided [0.015 to 0.285], Standard Deviation 0.069
Statistical Analysis 5: Comparison: Phase II GBM; 1-year progression free survival (n=21); Test type: Superiority or Other; Kaplan-Meier = 0.190, 95% CI 2-sided [0.039 to 0.341], Standard Deviation 0.077
Statistical Analysis 6: Comparison: Phase II GBM; 2-year progression free survival (n=21); Test type: Superiority or Other; Kaplan-Meier = 0.190, 95% CI 2-sided [0.039 to 0.341], Standard Deviation 0.077

8. Secondary Outcome: Ability of Erlotinib to Inhibit EGFR Signaling
Description: The objective was to test the ability of erlotinib to inhibit the EGFR signaling in patients with high-grade glioma who required a second surgery.
  This outcome was not assessed due to insufficient availability of tumor and control samples for analysis.
Time Frame: 5 Years
Population: This outcome was not assessed due to insufficient availability of tumor and control samples for analysis.
Groups:
- Patients With High-Grade/Low-Grade Glioma: Participants included patients with newly diagnosed high-grade glioma (excluding those originating in the brain stem) and unfavorable low-grade glioma who are ≥ 3 years and <26 years of age. Patients receiving enzyme-inducing anticonvulsants (EIACs) were not eligible for this study.
  Patients received erlotinib hydrochloride: In the Phase II component of this study, erlotinib was given at the MTD during and after RT for 2 years. The recommended dose of erlotinib for the Phase II component of the current study was 120mg/m^2 per day (maximum dose of 200mg per day).
Arm/Group | Patients With High-Grade/Low-Grade Glioma
Number analyzed (Participants) | 0

9. Secondary Outcome: Correlation Between Standard Magnetic Resonance Imaging and Investigational Radiologic Techniques in Assessing Tumor Response to This Treatment
Description: This objective was to prospectively investigate the correlation between standard magnetic resonance imaging (MRI) and investigational radiologic techniques (MR spectroscopy, perfusion/diffusion, PET scan, DEMRI/BLAST) in assessing tumor response to this treatment.
Time Frame: at diagnosis and regular intervals during therapy (up to 2 years after start of therapy)
Population: This objective became obsolete over the course of the protocol, and data was not collected.
Arm/Group | Patients With High-Grade/Low-Grade Glioma
Number analyzed (Participants) | 0

10. Secondary Outcome: To Prospectively Investigate the Technical Factors Involved in Planning and Administering Conformal Fractionated RT as Outlined in This Study, and to Correlate RT Dosimetry With Patterns of Failure, Standard and Investigational Imaging and Toxicity
Time Frame: 5 Years
Population: This objective became obsolete over the course of the protocol, and data was not collected.
Groups:
- Patients With High-Grade/Low-Grade Glioma: Patients with newly diagnosed high-grade glioma (excluding those originating in the brain stem) and unfavorable low-grade glioma who are ≥ 3 years and <26 years of age. Patients receiving enzyme-inducing anticonvulsants (EIACs) are not eligible for this study. Patients with spinal cord tumors will be eligible for the Phase I and Phase II component of this study, but they will not be taken into consideration to estimate PFS in the Phase II component of this trial because of their notoriously worse prognosis. Patients receive erlotinib hydrochloride.
  Erlotinib hydrochloride: This study had 2 components: a Phase I component which estimated the MTD and DLT(s) of erlotinib given once a day during and after conventionally fractionated RT for a period of 8 weeks (DLT-evaluation period), followed by continuous administration of this medication for up to 3 years; and a Phase II component where erlotinib was given at the MTD during and after RT for 2 years.
Arm/Group | Patients With High-Grade/Low-Grade Glioma
Number analyzed (Participants) | 0

11. Secondary Outcome: Plasma and CSF Levels of VEGF, bFGF, and SDF1
Description: This objective was to determine the plasma and CSF levels of the VEGF, bFGF, and SDF1 at diagnosis, and the plasma levels of these factors at regular intervals during therapy, and to analyze the association of these results with tumor response.
Time Frame: at diagnosis and regular intervals during therapy (up to 2 years after start of therapy)
Population: This objective became obsolete over the course of the protocol, and data was not collected.
Arm/Group | Patients With High-Grade/Low-Grade Glioma
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants Experiencing Grade 3 or 4 Toxicity Events
Description: Adverse events were collected systematically for each of the 44 Phase II participants from the time of enrollment to the completion of therapy (approximately 2 years from start of therapy).
Time Frame: From start of therapy through 2 years.
Population: All 44 Phase II participants were evaluated. Eight of 16 participants with lymphopenia received dexamethasone within 4 weeks of the recorded toxicity. In both participants with headache, there was a documented progressive disease within 3 days of the recorded headache.
Measure: Number; unit: Participants
Groups:
- Grade 3 Toxicity: Grade 3 toxicity per CTCAE 3.0.
- Grade 4 Toxicity: Grade 4 toxicity per CTCAE 3.0.
Arm/Group | Grade 3 Toxicity | Grade 4 Toxicity
Number analyzed (Participants) | 44 | 44
Participants
  Blood: Hemoglobin | 2 | 1
  Blood: Lymphopenia | 7 | 8
  Blood: Neutrophils | 2 | 1
  Blood: Platelets | 0 | 1
  Dermatologic: Pruritus | 3 | 0
  Dermatologic: Rash/Desquamation | 1 | 0
  Dermatologic: Rash/acne | 2 | 0
  Gastrointestinal: Anorexia | 3 | 0
  Gastrointestinal: Diarrhea | 5 | 0
  Gastrointestinal: Dysphagia | 1 | 0
  Gastrointestinal: Mucositis | 1 | 0
  Gastrointestinal: Nausea | 2 | 0
  Gastrointestinal: Vomiting | 4 | 0
  Metabolic: ALT/AST | 2 | 0
  Metabolic: Hypokalemia | 2 | 0
  Metabolic: Bilirubin | 1 | 0
  Pain: Headache | 1 | 1
  Constitutional: Fatigue | 1 | 0
  Constitutional: Weight Loss | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected systematically for each of the 23 Phase I and 44 Phase II participants from the time of enrollment to the completion of therapy (approximately 2 years from start of therapy).
Groups:
- 70 mg/m^2 (Phase I): Participants received dose of 70 mg/m^2, range of actual dose was 68-83 mg/m^2.
- 90 mg/m^2 (Phase I): Participants received dose of 90 mg/m^2, range of actual dose was 85-87.5 mg/m^2.
- 120 mg/m^2 (Phase I): Participants received dose of 120 mg/m^2, range of actual dose was 107-128 mg/m^2.
- 160 mg/m^2 (Phase I): Participants received dose of 160 mg/m^2, range of actual dose was 151.5-167 mg/m^2.
- Phase II: Phase II participants received 120 mg/m^2.
Arm/Group | 70 mg/m^2 (Phase I) | 90 mg/m^2 (Phase I) | 120 mg/m^2 (Phase I) | 160 mg/m^2 (Phase I) | Phase II
Serious Adverse Events (participants affected / at risk) | 4/7 | 1/3 | 2/7 | 4/6 | 26/44
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 7/7 | 6/6 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 70 mg/m^2 (Phase I) (N=7) | 90 mg/m^2 (Phase I) (N=3) | 120 mg/m^2 (Phase I) (N=7) | 160 mg/m^2 (Phase I) (N=6) | Phase II (N=44)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2) | 4 (6) | 16 (32) — Eight of the 16 patients with lymphopenia received dexamethasone within 4 weeks of the recorded toxicity.
Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash/Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
ALT/AST (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (4)
Bilirubin (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — There was a documented progressive disease within 3 days of the recorded headache.
Lipase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 70 mg/m^2 (Phase I) (N=7) | 90 mg/m^2 (Phase I) (N=3) | 120 mg/m^2 (Phase I) (N=7) | 160 mg/m^2 (Phase I) (N=6) | Phase II (N=44)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 8 (11)
Hearing: patients wihtout baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1 (4) | 2 (4) | 1 (1) | 0 (0) | 5 (6)
Hemoglobin (Blood and lymphatic system disorders) | 6 (15) | 2 (2) | 3 (3) | 4 (7) | 18 (41)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (10) | 2 (3) | 5 (6) | 3 (8) | 21 (38)
Lymphopenia (Blood and lymphatic system disorders) | 7 (18) | 3 (8) | 7 (14) | 6 (13) | 27 (104)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (6) | 1 (1) | 1 (1) | 1 (1) | 10 (16)
Platelets (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (3) | 3 (5) | 8 (10)
Supraventricular and nodal arrhythmia, sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 3 (4)
Hypertension (Cardiac disorders) | 3 (4) | 2 (2) | 2 (2) | 1 (1) | 6 (7)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (8) | 0 (0) | 2 (3) | 3 (4) | 18 (25)
Fever (in absence of neutrophenia defined as ANC <1.0 x 10e9/L) (General disorders) | 5 (8) | 1 (1) | 2 (2) | 1 (1) | 8 (10)
Insomnia (General disorders) | 1 (3) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Weight loss (General disorders) | 3 (4) | 0 (0) | 1 (1) | 2 (4) | 19 (27)
Chelitis (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Dermatology/Skin - other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 8 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (2) | 2 (2) | 4 (5) | 18 (19)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2) | 2 (3) | 1 (1) | 13 (14)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 7 (7)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (3) | 1 (1) | 16 (21)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2) | 4 (5) | 3 (4) | 19 (27)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 6 (8) | 3 (4) | 5 (5) | 2 (2) | 18 (29)
Striae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Cushingoid appearance(e.g. moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Anorexia (Gastrointestinal disorders) | 4 (10) | 2 (3) | 2 (3) | 5 (5) | 26 (30)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1) | 4 (4) | 8 (11)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 6 (13) | 3 (4) | 7 (8) | 4 (8) | 28 (51)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 8 (12)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 5 (5)
Mucositis/stomatitis (clinical exam), oral cavity (Gastrointestinal disorders) | 1 (1) | 3 (5) | 3 (3) | 1 (1) | 4 (4)
Mucositis/stomatitis (functional/symptomatic), oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (11) | 2 (5) | 3 (4) | 4 (6) | 19 (27)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (7)
Vomiting (Gastrointestinal disorders) | 5 (13) | 1 (3) | 3 (4) | 4 (5) | 19 (31)
Hemorrhage, pulmonary/upper respiratory, nose (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (6)
Infection - Other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 19 (26)
Infection with normal ANC or Grade 1 or 2 neurophils, external ear (otitis externa) (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils, middle ear (otitis media) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils, upper airway NOS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Opportunistic infection associated with >=Grade 2 lymphopenia (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 5 (6)
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2) | 3 (6) | 3 (3) | 2 (6) | 14 (26)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (5) | 13 (20)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 2 (2) | 1 (1) | 11 (19)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (6)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 4 (8) | 2 (5) | 16 (25)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (2) | 7 (12)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 4 (7)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6 (13) | 2 (2) | 1 (1) | 3 (5) | 13 (23)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (3) | 8 (14)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (13) | 4 (5) | 9 (15)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (10) | 2 (7) | 2 (3) | 4 (5) | 12 (22)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (10) | 0 (0) | 2 (3) | 3 (5) | 12 (23)
Musculoskeletal/soft tissue - other (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Ataxia (incoordination) (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 8 (13)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 3 (3)
Mood alteration, anxiety (Nervous system disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Mood alteration, depression (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 6 (8)
Neurology - other (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (12)
Neuropathy: motor (Nervous system disorders) | 3 (7) | 0 (0) | 3 (3) | 4 (4) | 4 (6)
Seizure (Nervous system disorders) | 3 (4) | 1 (1) | 4 (4) | 3 (3) | 11 (25)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Nystagmus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ocular/visual - other (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 10 (11)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Vision-blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 2 (2) | 1 (1) | 2 (4) | 7 (7)
Pain - other (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 11 (17)
Pain, abdomen NOS (General disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (3) | 6 (7)
Pain, back (General disorders) | 1 (2) | 1 (2) | 2 (2) | 1 (1) | 4 (5)
Pain, head/headache (General disorders) | 5 (17) | 2 (3) | 3 (4) | 5 (6) | 20 (29)
Pain, throat/pharynx/larynx (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 7 (7)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 3 (4)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 4 (10) | 1 (4) | 15 (28)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Auditory/Ear - other (Ear and labyrinth disorders) | 5 (8) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Otitis, middle ear (non-infectious (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rigors/chills (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
Dental: teeth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hemorrhage, CNS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hemorrhage, GU, urinary NOS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, Anal/perianal (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, eye NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, mucosa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, pharynx (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, sinus (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, skin (cellulitis) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, urinary tract NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, wound (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Personality/behavioral (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular surface disease (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
Vision-photophobia (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain, chest/thorax NOS (General disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Pain, external ear (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain, eye (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain, joint (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 2 (3)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils, lip/perioral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Supraventricular and nodal arrhythmia, sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight gain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash: dermatitis associated with radiation, radiation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Death not associated with CTCAE term, disease progression NOS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Death occurred due to a sledding accident. Participant had completed all therapy and was in follow-up.
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (including bile reflex gastritis) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ulcer, GI, stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary/pancreas - other (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, conjunctiva (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, dental-tooth (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, Foreign body (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — e.g., graft, implant, prosthesis, stent
Infection with normal ANC or Grade 1 or 2 neutrophils, lung (pnemonia) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils, meninges (meningitis) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, nose (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, oral cavity-gums (gingivitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, rectum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholesterol, serum-high (hypercholestremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metabolic/laboratory - other (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy), whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trismus (difficulty, restriction or pain when opening mouth) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leak, cerebrospinal fluid (CSF) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood alteration, agitation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neuropathy: cranial, CN VI Lateral deviation of eye (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy: cranial, CN VII motor-face: sensory-taste (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy: cranial, CN VIII hearing and balance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyramidal tract dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — (e.g., increased tone, hyperreflexia, positive Babinski, decreased motor coordination)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid dysfunction (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary/upper respiratory - other (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Secondary malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sexual/reproductive function - other (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-operative injury, brain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flu-like syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain, extremity-limb (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain, muscle (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain, oral cavity (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain, pain NOS (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain, stomach (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Lymphatics - other (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes